CLINICAL TRIAL: NCT04752930
Title: Circulating Tumor DNA (ctDNA) as a Assisted Diagnosis, Early Intervention and Prognostic Marker for Peritoneal Metastases From Colorectal Cancer: A Prospective, Open-label, Randomized Controlled Study
Brief Title: ctDNA as a Assisted Diagnosis, Early Intervention and Prognostic Marker for Peritoneal Metastases From Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SixthSunYetSen-ctDNA
Record Dates: First submitted 2021-01-26; First posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-01

CONDITIONS: Colorectal Cancer; Peritoneal Metastases
Keywords: ctDNA
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ctDNA monitoring (Experimental): ctDNA monitoring will be performed at protocol-specified intervals and requirement
  Interventions: Diagnostic Test: ctDNA monitoring
- Imageology (SOC) (Active Comparator): Imaging examination will be performed at protocol-specified intervals and requirement
  Interventions: Diagnostic Test: Imageology

INTERVENTIONS:
Diagnostic Test: ctDNA monitoring — Patients who undergoing radical surgery for colorectal cancer for 6~12 months and with 2 consecutive positive ctDNA testing results within 1 month will be enrolled, and diagnostic laparoscopy will be performed immediately after enrollment. Patients with positive peritoneal metastasis (PCI score <20) will be treated with CRS+HIPEC. Tumor markers, endoscopic and imaging examinations, and ctDNA monitoring will be performed every 3 months in patients with negative peritoneal metastasis. Laparoscopy will be performed when imaging suggested peritoneal metastasis (oligometastases). Re-diagnostic laparoscopy will be performed 24 months after radical surgery when there is no radiographic evidence of recurrence or metastasis. Follow-up time will up to 36 months after colorectal cancer surgery.
  Arms: ctDNA monitoring
Diagnostic Test: Imageology — Patients who undergoing radical surgery for colorectal cancer for 6~12 months and with 2 consecutive positive ctDNA testing results within 1 month will be enrolled. and there will be no need to conduct endoscopic exploration immediately after enrollment. Tumor markers, endoscopic and imaging examinations, and ctDNA monitoring will be performed every 3 months until imaging suggested peritoneal metastasis (oligometastases). Patients with positive peritoneal metastasis (PCI score <20) will be treated with CRS+HIPEC. Re-diagnostic laparoscopy will be performed 24 months after radical surgery when there is no radiographic evidence of recurrence or metastasis. Follow-up time will up to 36 months after colorectal cancer surgery.
  Arms: Imageology (SOC)

SUMMARY:
This is a prospective, open-label, randomized controlled clinical trial, by monitoring the serum ctDNA mutational profile using NGS, aiming to elucidate the correlation between the postoperative ctDNA status and the assisted diagnosis, early intervention and prognosis for colorectal cancer peritoneal metastases.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be a man or woman of at 18-75;
* Patients must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-21；
* Patients with primary colorectal cancer proven by pathology；
* Patients with high risk factors for peritoneal metastasis (simultaneous peritoneal metastasis, ovarian metastasis, PT4, CT4, tumor perforation, tumor-complete intestinal obstruction, mucinous adenocarcinoma/signet ring cell carcinoma of PT3, positive surgical margin, and tumor rupture and hemorrhage);
* 6-12 months after colorectal cancer radical surgery, patients who have two consecutive positive ctDNA tests within one month;
* Patients who have finished standard adjuvant therapy after surgery; (Choose 5-FU or 5-FU analog-based chemotherapy regimen, and the perioperative chemotherapy should not exceed 6 months)；
* Patients who are negative of recurrence or metastasis in conventional oncology examination (serology, endoscopy, imaging) ;
* Written informed consent must be obtained from patients and ability for patients to comply with the requirements of the study.

Exclusion Criteria:

* Patients who were diagnosed with other malignant tumors within 2 years before diagnosis of colorectal cancer;
* ASA class Ⅳ to Ⅴ;
* Patients who have other existence of distant metastasis outside the abdomen;
* Patients with serious mental illness;
* Patients with severe cardiovascular disease, uncontrollable infections, or other uncontrollable co-diseases;
* Patients who cannot be followed up as scheduled;
* Patients who participated in other clinical studies within 3 months prior to the trial;
* Pregnant or nursing women, men or women of childbearing potential who are unwilling to employ adequate contraception.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2020-08-24 (Actual); Primary Completion 2023-09-24 (Estimated); Study Completion 2025-08-24 (Estimated)

PRIMARY OUTCOMES:
Peritoneal Metastasis Free Survival (PMFS) | Through study completion, up to 3 years
  The survival rate without peritoneal metastasis (oligometastatic) at 24 months after radical resection of colorectal cancer.

SECONDARY OUTCOMES:
Detection Rate (DR) | Interim analyses: After 69 patients have been enrolled, up to 1.5 years
  DR of ctDNA monitoring for predicting peritoneal metastasis with abdominal exploration as the reference.
  DR of imageological examination for predicting peritoneal metastasis with abdominal exploration as the reference.
  DR of combination of ctDNA monitoring and imageological examination for predicting peritoneal metastasis with abdominal exploration as the reference.
  Will be compared in both arms.
Positive Percent Agreement (PPA) | Interim analyses: After 69 patients have been enrolled, up to 1.5 years
  PPA of ctDNA monitoring for predicting peritoneal metastasis with abdominal exploration as the reference.
  PPA of imageological examination for predicting peritoneal metastasis with abdominal exploration as the reference.
  PPA of combination of ctDNA monitoring and imageological examination for predicting peritoneal metastasis with abdominal exploration as the reference.
  Will be compared in both arms.
Negative Percent Agreement (NPA) | Interim analyses: After 69 patients have been enrolled, up to 1.5 years
  NPA of ctDNA monitoring for predicting peritoneal metastasis with abdominal exploration as the reference.
  NPA of imageological examination for predicting peritoneal metastasis with abdominal exploration as the reference.
  NPA of combination of ctDNA monitoring and imageological examination for predicting peritoneal metastasis with abdominal exploration as the reference.
  Will be compared in both arms.
The time of peritoneal metastasis diagnosed after radical surgery | Interim analyses: After 69 patients have been enrolled, up to 1.5 years
  Will be compared in both arms.
Peritoneal Cancer Index (PCI) Score | Interim analyses: After 69 patients have been enrolled, up to 1.5 years
  This scale measures the extent of peritoneal cancer throughout the peritoneal cavity.
  The range of this scale is from 0 to 39.
  0 = no disease within the peritoneal cavity
  0-9 = minimal disease
  10-29 = moderate disease
  30-39 = extensive disease
  Lower values are considered a better outcome for the patient.
  Will be compared in both arms.
Completeness of Cytoreduction (CC) Score | Interim analyses: After 69 patients have been enrolled, up to 1.5 years
  The degree to which the disease was able to be excised during the procedure.
  This scale ranges from CC0-CC3.
  CC0 = all disease has been cleared, with no visible peritoneal carcinomatosis after CRS
  CC1 = microscopic disease remains (Nodules persisting < 2.5 mm after CRS)
  CC2 = macroscopic disease remains (Nodules persisting between 2.5 mm and 2.5 cm)
  CC3 = Substantial Macroscopic disease remains (Nodules persisting > 2.5 cm)
  Lower values are considered a better outcome, with CC0/1 classed as favourable and CC2/3 indicating an incomplete clearance of disease.
  Will be compared in both arms.
The ctDNA clearance rate before and after CRS+HIPEC treatment | Interim analyses: After 69 patients have been enrolled, up to 1.5 years
  Will be compared in both arms.
The rate of Disease Free Survival (DFS) at 3 years after radical resection of colorectal cancer | Through study completion, up to 3 years
  Whether the patient is still alive and free of disease or not.
  Will be compared in both arms.
The Overall Survival (OS) at 3 years after radical resection of colorectal cancer | Through study completion, up to 3 years
  Whether the patient is still alive or not.
  Will be compared in both arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Franko J, Shi Q, Goldman CD, Pockaj BA, Nelson GD, Goldberg RM, Pitot HC, Grothey A, Alberts SR, Sargent DJ. Treatment of colorectal peritoneal carcinomatosis with systemic chemotherapy: a pooled analysis of north central cancer treatment group phase III trials N9741 and N9841. J Clin Oncol. 2012 Jan 20;30(3):263-7. doi: 10.1200/JCO.2011.37.1039. Epub 2011 Dec 12. PMID 22162570
- [Background] Yonemura Y, Bandou E, Kawamura T, Endou Y, Sasaki T. Quantitative prognostic indicators of peritoneal dissemination of gastric cancer. Eur J Surg Oncol. 2006 Aug;32(6):602-6. doi: 10.1016/j.ejso.2006.03.003. Epub 2006 Apr 17. PMID 16617004
- [Background] Elias D, Lefevre JH, Chevalier J, Brouquet A, Marchal F, Classe JM, Ferron G, Guilloit JM, Meeus P, Goere D, Bonastre J. Complete cytoreductive surgery plus intraperitoneal chemohyperthermia with oxaliplatin for peritoneal carcinomatosis of colorectal origin. J Clin Oncol. 2009 Feb 10;27(5):681-5. doi: 10.1200/JCO.2008.19.7160. Epub 2008 Dec 22. PMID 19103728
- [Background] Baratti D, Kusamura S, Deraco M. The Fifth International Workshop on Peritoneal Surface Malignancy (Milan, Italy, December 4-6, 2006): methodology of disease-specific consensus. J Surg Oncol. 2008 Sep 15;98(4):258-62. doi: 10.1002/jso.21056. PMID 18726888
- [Background] Esquivel J, Chua TC, Stojadinovic A, Melero JT, Levine EA, Gutman M, Howard R, Piso P, Nissan A, Gomez-Portilla A, Gonzalez-Bayon L, Gonzalez-Moreno S, Shen P, Stewart JH, Sugarbaker PH, Barone RM, Hoefer R, Morris DL, Sardi A, Sticca RP. Accuracy and clinical relevance of computed tomography scan interpretation of peritoneal cancer index in colorectal cancer peritoneal carcinomatosis: a multi-institutional study. J Surg Oncol. 2010 Nov 1;102(6):565-70. doi: 10.1002/jso.21601. PMID 20976729
- [Background] Dromain C, Leboulleux S, Auperin A, Goere D, Malka D, Lumbroso J, Schumberger M, Sigal R, Elias D. Staging of peritoneal carcinomatosis: enhanced CT vs. PET/CT. Abdom Imaging. 2008 Jan-Feb;33(1):87-93. doi: 10.1007/s00261-007-9211-7. PMID 17632751
- [Background] Bettegowda C, Sausen M, Leary RJ, Kinde I, Wang Y, Agrawal N, Bartlett BR, Wang H, Luber B, Alani RM, Antonarakis ES, Azad NS, Bardelli A, Brem H, Cameron JL, Lee CC, Fecher LA, Gallia GL, Gibbs P, Le D, Giuntoli RL, Goggins M, Hogarty MD, Holdhoff M, Hong SM, Jiao Y, Juhl HH, Kim JJ, Siravegna G, Laheru DA, Lauricella C, Lim M, Lipson EJ, Marie SK, Netto GJ, Oliner KS, Olivi A, Olsson L, Riggins GJ, Sartore-Bianchi A, Schmidt K, Shih lM, Oba-Shinjo SM, Siena S, Theodorescu D, Tie J, Harkins TT, Veronese S, Wang TL, Weingart JD, Wolfgang CL, Wood LD, Xing D, Hruban RH, Wu J, Allen PJ, Schmidt CM, Choti MA, Velculescu VE, Kinzler KW, Vogelstein B, Papadopoulos N, Diaz LA Jr. Detection of circulating tumor DNA in early- and late-stage human malignancies. Sci Transl Med. 2014 Feb 19;6(224):224ra24. doi: 10.1126/scitranslmed.3007094. PMID 24553385
- [Background] Abbosh C, Birkbak NJ, Wilson GA, Jamal-Hanjani M, Constantin T, Salari R, Le Quesne J, Moore DA, Veeriah S, Rosenthal R, Marafioti T, Kirkizlar E, Watkins TBK, McGranahan N, Ward S, Martinson L, Riley J, Fraioli F, Al Bakir M, Gronroos E, Zambrana F, Endozo R, Bi WL, Fennessy FM, Sponer N, Johnson D, Laycock J, Shafi S, Czyzewska-Khan J, Rowan A, Chambers T, Matthews N, Turajlic S, Hiley C, Lee SM, Forster MD, Ahmad T, Falzon M, Borg E, Lawrence D, Hayward M, Kolvekar S, Panagiotopoulos N, Janes SM, Thakrar R, Ahmed A, Blackhall F, Summers Y, Hafez D, Naik A, Ganguly A, Kareht S, Shah R, Joseph L, Marie Quinn A, Crosbie PA, Naidu B, Middleton G, Langman G, Trotter S, Nicolson M, Remmen H, Kerr K, Chetty M, Gomersall L, Fennell DA, Nakas A, Rathinam S, Anand G, Khan S, Russell P, Ezhil V, Ismail B, Irvin-Sellers M, Prakash V, Lester JF, Kornaszewska M, Attanoos R, Adams H, Davies H, Oukrif D, Akarca AU, Hartley JA, Lowe HL, Lock S, Iles N, Bell H, Ngai Y, Elgar G, Szallasi Z, Schwarz RF, Herrero J, Stewart A, Quezada SA, Peggs KS, Van Loo P, Dive C, Lin CJ, Rabinowitz M, Aerts HJWL, Hackshaw A, Shaw JA, Zimmermann BG; TRACERx consortium; PEACE consortium; Swanton C. Phylogenetic ctDNA analysis depicts early-stage lung cancer evolution. Nature. 2017 Apr 26;545(7655):446-451. doi: 10.1038/nature22364. PMID 28445469
- [Background] Tie J, Wang Y, Tomasetti C, Li L, Springer S, Kinde I, Silliman N, Tacey M, Wong HL, Christie M, Kosmider S, Skinner I, Wong R, Steel M, Tran B, Desai J, Jones I, Haydon A, Hayes T, Price TJ, Strausberg RL, Diaz LA Jr, Papadopoulos N, Kinzler KW, Vogelstein B, Gibbs P. Circulating tumor DNA analysis detects minimal residual disease and predicts recurrence in patients with stage II colon cancer. Sci Transl Med. 2016 Jul 6;8(346):346ra92. doi: 10.1126/scitranslmed.aaf6219. PMID 27384348
- [Background] Saluja H, Karapetis CS, Pedersen SK, Young GP, Symonds EL. The Use of Circulating Tumor DNA for Prognosis of Gastrointestinal Cancers. Front Oncol. 2018 Jul 24;8:275. doi: 10.3389/fonc.2018.00275. eCollection 2018. PMID 30087854
- [Background] Ossandon MR, Agrawal L, Bernhard EJ, Conley BA, Dey SM, Divi RL, Guan P, Lively TG, McKee TC, Sorg BS, Tricoli JV. Circulating Tumor DNA Assays in Clinical Cancer Research. J Natl Cancer Inst. 2018 Sep 1;110(9):929-934. doi: 10.1093/jnci/djy105. PMID 29931312
- [Background] Yang QM, Bando E, Kawamura T, Tsukiyama G, Nemoto M, Yonemura Y, Furukawa H. The diagnostic value of PET-CT for peritoneal dissemination of abdominal malignancies. Gan To Kagaku Ryoho. 2006 Nov;33(12):1817-21. PMID 17212117
- [Background] Yonemura Y, Elnemr A, Endou Y, Hirano M, Mizumoto A, Takao N, Ichinose M, Miura M, Li Y. Multidisciplinary therapy for treatment of patients with peritoneal carcinomatosis from gastric cancer. World J Gastrointest Oncol. 2010 Feb 15;2(2):85-97. doi: 10.4251/wjgo.v2.i2.85. PMID 21160926
- [Background] Satoh Y, Ichikawa T, Motosugi U, Kimura K, Sou H, Sano K, Araki T. Diagnosis of peritoneal dissemination: comparison of 18F-FDG PET/CT, diffusion-weighted MRI, and contrast-enhanced MDCT. AJR Am J Roentgenol. 2011 Feb;196(2):447-53. doi: 10.2214/AJR.10.4687. PMID 21257899
- [Background] Brucher BL, Piso P, Verwaal V, Esquivel J, Derraco M, Yonemura Y, Gonzalez-Moreno S, Pelz J, Konigsrainer A, Strohlein M, Levine EA, Morris D, Bartlett D, Glehen O, Garofalo A, Nissan A. Peritoneal carcinomatosis: cytoreductive surgery and HIPEC--overview and basics. Cancer Invest. 2012 Mar;30(3):209-24. doi: 10.3109/07357907.2012.654871. PMID 22360361
- [Background] Koh JL, Yan TD, Glenn D, Morris DL. Evaluation of preoperative computed tomography in estimating peritoneal cancer index in colorectal peritoneal carcinomatosis. Ann Surg Oncol. 2009 Feb;16(2):327-33. doi: 10.1245/s10434-008-0234-2. Epub 2008 Dec 3. PMID 19050972
- [Background] Rausei S, Ruspi L, Mangano A, Lianos GD, Galli F, Boni L, Roukos DH, Dionigi G. Advantages of staging laparoscopy in gastric cancer: they are so obvious that they are not evident. Future Oncol. 2015;11(3):369-72. doi: 10.2217/fon.14.283. No abstract available. PMID 25675119
- [Background] Stroun M, Anker P, Maurice P, Lyautey J, Lederrey C, Beljanski M. Neoplastic characteristics of the DNA found in the plasma of cancer patients. Oncology. 1989;46(5):318-22. doi: 10.1159/000226740. PMID 2779946